CLINICAL TRIAL: NCT07267767
Title: Comparison of Six Different Machine Learning Methods With Traditional Model for Low Anterior Resection Syndrome After Minimally Invasive Surgery for Rectal Cancer -- Development and External Validation of a Nomogram : A Dual-center Cohort Study
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Collaborators: China-Japan Union Hospital, Jilin University (Other)
Responsible Party: Principal Investigator, Daorong Wang, NANJING UNIVERSITY, Northern Jiangsu People's Hospital
Other Study IDs: jiangsuNorthen20
Record Dates: First submitted 2025-07-09; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer; LARS - Low Anterior Resection Syndrome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Months

INTERVENTIONS:
Procedure: nCRT — neoadjuvant chemoradiotherapy
Behavioral: BMI — Body Mass Index
Diagnostic Test: Distance from AV — Distance from AV
Procedure: Surgical type — laparoscopic and robotic surgery
Procedure: Surgical approach — tatme + isr
Procedure: LCA Preserving — LCA Preserving
Procedure: Prophylactic stoma — Prophylactic stoma
Procedure: Anastomotic leakage — Anastomotic leakage

SUMMARY:
Following thorough screening based on inclusion and exclusion criteria, patients from the two sizable medical centers were split up into two cohorts for this study. Cohort 1 served primarily as the training and internal validation set, while Cohort 2 was used for external validation of the predictive model constructed from Cohort 1. We used six distinct machine learning methodss, including DT, RF, XGBOOST, SVM, lightGBM, and SHLNN, in addition to conventional logistic regression to create the predictive model. We chose the approach with the best sensitivity and specificity by comparing the concordance index(C-index) akin to the area under the ROC curve (AUC) of these seven distinct model-building methods. The predictive model for Cohort 1 was then built using this method, and internal validation was finished. Lastly, Cohort 2 underwent external validation of the predictive model

ELIGIBILITY:
Inclusion Criteria:(1) rectal adenocarcinoma (2) minimally invasive sphincter-preserving surgery (taTME/ISR/LAR) (3) intact baseline anal function (4) no emergent presentations or metastases.

-

Exclusion Criteria:emergent presentations or metastases

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective analysis included 3,937 radical rectal cancer cases from two Chinese university hospitals (Northern Jiangsu People's Hospital 2015-2023, n=2612; Jilin University's China-Japan Union Hospital 2021-2023, n=1325), with rigorous selection criteria ensuring cohort homogeneity
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
low anterior resection syndrome | 1 and 3 months after surgery
Comparison of Six Different Machine Learning Methods With Traditional Model for Low Anterior Resection Syndrome After Minimally Invasive Surgery for Rectal Cancer -- Development and External Validation of a Nomogram : A Dual-center Cohort Study | 3 months
  using LARS Score to assess the LARS situation